CLINICAL TRIAL: NCT04768439
Title: Comparison Between Low and High Doses of Prophylactic Vitamin D in Prevention of Osteopenia of Prematurity
Brief Title: Low and High Doses of Prophylactic Vitamin D in Prevention of Osteopenia of Prematurity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00007555-00015712
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Osteopenia of Prematurity
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Vitamin D; Calcitriol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 200 IU/d vitamin D (Experimental): Patients will receive low-dose vitamin D (200 IU/d)
  Interventions: Drug: Low Dose Vitamin D
- 1600 IU/d vitamin D (Experimental): Patients will receive high-dose vitamin D (1600 IU/d)
  Interventions: Drug: High Dose Vitamin D

INTERVENTIONS:
Drug: Low Dose Vitamin D — Patients will receive a 200 IU/d vitamin D since they tolerate full enteral nutrition.
  Other Names: 1,25-Dihydroxycholecalciferol
  Arms: 200 IU/d vitamin D
Drug: High Dose Vitamin D — Patients will receive 1600 IU/d vitamin D since they tolerate full enteral nutrition.
  Other Names: 1,25-Dihydroxycholecalciferol
  Arms: 1600 IU/d vitamin D

SUMMARY:
In this study the effects of low and high doses of prophylactic vitamin D on biochemical and radiological manifestations of osetopenia of prematurity will be tested.

DETAILED DESCRIPTION:
The study will be conducted on (80) preterm infants that fulfill the eligibility criteria and delivered at Alexandria University Maternity Hospital (AUMH).

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age of ≤ 32 weeks and birth weight ≤ 1500 g.

Exclusion Criteria:

* Newborns whose mothers were taking specific medications interacting with vitamin D metabolism (e.g., anticonvulsants, diuretics)
* Being NPO (nothing per oral) for more than 2 wks
* Gestational age more than 32 weeks
* Birth weight more than 1500 grams

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Calcium level and activity | six weeks
  Serum calcium level will be measured and analyzed using Advia 1800 chemistry system (Simens Germany). Normal level: 8.5 to 10.5 mg/dl
Phosphorus level and activity | six weeks
  Serum phosphorus level will be measured and analyzed using Advia 1800 chemistry system (Simens Germany). Normal level: 3.4 to 4.5 mg/dl
Alkaline phosphatase level and activity | six weeks
  Serum alkaline phosphate level will be measured and analyzed using Advia 1800 chemistry system (Simens Germany). Normal level: 50-100 U/L.
25-Hydroxy Vitamin D | six weeks
  Serum 25-Hydroxy Vitamin D level will be measured and analyzed using Electrochemilumiescence binding assay on cobas e immunoassay analyzer. The reference range of the total 25(OH)D level is 25-80 ng/mL.
Bone fracture | six weeks
  This will be evaluated using an x-ray of left wrist
Intracortical resorption | six weeks
  This will be evaluated using an x-ray of left wrist
Losing the sharp bone border (fraying) | six weeks
  This will be evaluated using an x-ray of left wrist
Cupping of metaphyseal edge of bone | six weeks
  This will be evaluated using an x-ray of left wrist
Widening of the distal end of the metaphysis of bone | six weeks
  This will be evaluated using an x-ray of left wrist

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Farrag, PhD, Principal Investigator — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt